CLINICAL TRIAL: NCT05307263
Title: Combination Therapy of Atherectomy Plus Drug-coated Balloon Versus Drug-coated Balloon for Complex Femoropopliteal Artery Disease (ARTEMIS Trial)
Brief Title: Combination Therapy of Atherectomy Plus Drug-coated Balloon Versus Drug-coated Balloon for Complex Femoropopliteal Artery Disease
Acronym: ARTEMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0051
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Femoropopliteal Artery Disease
Keywords: Femoropopliteal artery disease; drug-coated balloon; angioplasty; atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atherectomy plus DCB (Active Comparator)
  Interventions: Procedure: Combination therapy of atherectomy and DCB
- DCB (Active Comparator)
  Interventions: Procedure: DCB alone

INTERVENTIONS:
Procedure: Combination therapy of atherectomy and DCB — The target lesion in femoropopliteal artery will be treated with atherectomy folloewd by DCB. The choice of atherectomy devices (HawkOne, Jectstream, or Rotarex)and DCBs (IN.PACT or Ranger) will be left to the operator's decision. In presence of ≥ 50% residual stenosis or flow limiting dissections, implantation of bare nitinol stents is recommended. Implantational of drug-eluting stents is not allowed.
  Arms: Atherectomy plus DCB
Procedure: DCB alone — The target lesion in femoropopliteal artery will be treated with DCB. The choice of DCBs (IN.PACT or Ranger) will be left to the operator's decision. In presence of ≥ 50% residual stenosis or flow limiting dissections, implantation of bare nitinol stents is recommended. Implantational of drug-eluting stents is not allowed.
  Arms: DCB

SUMMARY:
* Prospective, multi-center, randomized, controlled comparison study
* A total of 300 subjects with complex femoropopliteal artery disease will be included according to inclusion and exclusion criteria. Complex lesions include long lesions (>150 mm), calcified lesions (PACSS grade 2-4) and in-stent lesions.
* Patients will be randomized in a 1:1 manner into atherectomy plus drug-coated balloon (DCB) or angiography-guided intervention group. • The randomization will be startified by the participating center and in-stent restenosis lesion. • For the DCB treatment, either IN.PACT (Medtronic) or Ranger (Boston Scientific) DCB will be used. • For the atherectomy, HawkOne (Medtronic), Jetstream (Boston scientific), or Rotarex (Straub Medical) will be used. • The primary endpoint is primary patency at 12 months based on Kaplan-Meier survival analysis. • Ankle-brachial index and Image study follow-up (Duplex US, CT angiography, or catheter angiography) will be performed at 1 year.
* Patients will be followed clinically for 2 years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Symptomatic peripheral artery disease:

   * Moderate or severe claudication (Rutherford category 2 or 3)
   * Critical limb ischemia (Rutherford category 4 or 5)
3. Femoropopliteal artery disease (stenosis > 50%) with one of following complex lesion characteristics: - long lesion (>150 mm), in-stent restenosis, calcified lesion (PACCS grade 2-4)
4. Femoropopliteal artery lesions that operators consider appropriate for treatment with both atherectomy plus drug-coated balloons and drug-coated balloons alone
5. Patients with signed informed consent

Exclusion Criteria:

1. Acute critical limb ischemia
2. Severe critical limb ischemia (Rutherford category 6)
3. Contraindication to any of the following medications: heparin, aspirin, clopidogrel, or contrast agents due to severe hypersensitive reactions
4. Age > 85 years
5. Severe hepatic dysfunction (> 3 times normal reference values)
6. Significant thrombocytopenia, anemia, or known bleeding diathesis
7. LVEF < 35% or clinically overt congestive heart failure
8. Pregnant women or women with potential childbearing
9. Life expectancy <1 year due to comorbidity
10. Previous bypass surgery in the target femoropopliteal artery
11. Untreated inflow disease of the ipsilateral pelvic or femoropopliteal arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months post treatment
  Primary patency is defined as absence of restenosis >50% by Duplex ultrasound, CT angiography, or catheter-based angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No